CLINICAL TRIAL: NCT06910254
Title: Effects of Overground Robot-Assisted Gait Training and Recumbent Bicycle Training on Muscle Characteristics, Falls Efficacy, and Physical Function in Patients With Subacute Stroke-Related Sarcopenia
Brief Title: Effects of Overground Robot-Assisted Gait Training on Stroke-Related Sarcopenia
Acronym: oRAGT-PSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Dong min park, Principal Investigator, Clinical physical therapist, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2025-01-010-004
Record Dates: First submitted 2025-03-17; First posted 2025-04-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Sarcopenia; Muscle Atrophy; Mobility Limitation; Muscle Quality; Robotic Rehabilitation
Keywords: subacute stroke; sarcopenia; Overground Robot-Assisted Gait Training (o-RAGT); Robotic rehabilitation; Muscle Quality; Skeletal muscle mass; Falls Efficacy; Exoskeleton Robot
MeSH Terms: conditions — Stroke; Sarcopenia; Muscular Atrophy; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: This study is a single-center, randomized controlled trial with a two-arm parallel-group design. A total of 53 participants with subacute stroke-related sarcopenia were randomly assigned to either an experimental group or a control group. Both groups received a 4-week intervention consisting of five 60-minute sessions per week.
  Participants in the experimental group received 30 minutes of overground robot-assisted gait training (o-RAGT) using the Angel Legs M20 exoskeleton, followed by 30 minutes of recumbent bicycle (RC) training. Participants in the control group received 60 minutes of recumbent bicycle training alone.
  Per-protocol analyses were conducted for participants who completed the full intervention and outcome assessments, resulting in a final sample of 41 participants (experimental group, n=19; control group, n=22).
Who Masked: Outcomes Assessor
Masking Description: This study employed a single-blind design. Due to the nature of the interventions, participants and therapists delivering the overground robot-assisted gait training and recumbent bicycle training could not be blinded to group allocation.
  However, outcome assessors were blinded to group assignments throughout the study. All primary and secondary outcome assessments were performed by assessors who were not involved in the intervention delivery and had no access to the randomization information during data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- o-RAGT + Recumbent Bicycle Training (Experimental): Participants in the experimental group received a combined intervention consisting of 30 minutes of overground robot-assisted gait training (o-RAGT) followed by 30 minutes of recumbent bicycle (RC) training. The o-RAGT was performed using the Angel Legs M20 wearable exoskeleton. The intervention was conducted five sessions per week for a total of 4 weeks (20 sessions).
  Interventions: Device: Overground Robot-Assisted Gait Training (o-RAGT); Device: Recumbent Bicycle Training
- Recumbent Bicycle Training Only (Active Comparator): Participants in the control group received 60 minutes of recumbent bicycle (RC) training alone to match the total exercise duration of the experimental group. The training was conducted five sessions per week for a total of 4 weeks (20 sessions).
  Interventions: Device: Recumbent Bicycle Training

INTERVENTIONS:
Device: Overground Robot-Assisted Gait Training (o-RAGT) — This intervention consists of overground robot-assisted gait training (o-RAGT) performed using the Angel Legs M20 wearable exoskeleton (Angel Robotics, Seoul, Republic of Korea). Participants perform structured overground walking practice with robotic assistance during scheduled training sessions. The device is used to support repetitive, task-specific overground gait practice under supervised clinical conditions.
  Other Names: Angel Legs M20 wearable exoskeleton
  Arms: o-RAGT + Recumbent Bicycle Training
Device: Recumbent Bicycle Training — Participants perform recumbent bicycle training using a stationary recumbent cycle ergometer (DRAX TBR9000, Republic of Korea). Training is conducted in a seated position with lower-extremity pedaling at a prescribed intensity. Each session is performed according to the study protocol under supervised clinical conditions.
  Other Names: Recumbent ergometer

SUMMARY:
This single-center randomized controlled trial evaluates the effects of combining overground robot-assisted gait training (o-RAGT) with recumbent cycling (RC) compared with RC alone in patients with subacute stroke at risk of sarcopenia. The study examines changes in muscle characteristics (muscle mass and quality), falls efficacy, and physical function following a 4-week intervention. Participants are randomly assigned to receive either combined o-RAGT and RC or RC alone. The findings aim to inform the potential role of overground robot-assisted gait training as an adjunctive intervention in stroke rehabilitation.

DETAILED DESCRIPTION:
This study is a single-center, randomized controlled trial designed to evaluate the effects of combining overground robot-assisted gait training (o-RAGT) with recumbent cycling (RC) in patients with subacute stroke at risk of sarcopenia. A total of 53 participants were randomly assigned to either an experimental group receiving combined o-RAGT and RC or a control group receiving RC alone.

The intervention was conducted five times per week for 60 minutes per session over a 4-week period. Overground robot-assisted gait training was performed using the Angel Legs M20 exoskeleton, while recumbent cycling was provided as conventional exercise training.

The primary outcomes were changes in skeletal muscle mass index, muscle quality, and falls efficacy. Secondary outcomes included measures of physical performance and functional mobility, such as the Short Physical Performance Battery, 6-Minute Walk Test, Timed Up and Go test, and lower extremity motor function.

This study aims to provide clinical information regarding the feasibility and potential effects of combining overground robot-assisted gait training with conventional exercise in stroke rehabilitation.

ELIGIBILITY:
- Inclusion Criteria

Participants must meet all of the following criteria:

1. Diagnosis of stroke within 6 months of onset (subacute phase), corresponding to the active neurological recovery period.
2. Classified as having possible sarcopenia according to the Asian Working Group for Sarcopenia (AWGS 2019) algorithm, defined by:

   * A positive SARC-F screening, and
   * Either reduced handgrip strength (men <28 kg, women <18 kg) or reduced physical performance (SPPB score <9).
3. Height between 140 and 190 cm and body weight ≤80 kg, meeting the mechanical fitting requirements of the overground wearable gait robot used in this study.
4. Functional Ambulation Category (FAC) score ≥1, indicating the ability to attempt ambulation with at least minimal assistance.
5. Korean version of the Mini-Mental State Examination (MMSE-K) score ≥24, indicating sufficient cognitive ability to understand instructions and participate in training.
6. Currently admitted for inpatient rehabilitation at a rehabilitation hospital in Seoul, Republic of Korea.
7. Ability and willingness to provide written informed consent after receiving a full explanation of the study procedures, potential risks, and benefits.

   * Exclusion Criteria

Participants will be excluded if they meet any of the following criteria:

1. Presence of severe cardiovascular disease (e.g., unstable angina, heart failure, recent myocardial infarction) or acute medical infection that contraindicates exercise-based interventions.
2. Musculoskeletal conditions that preclude safe participation in robotic gait training or recumbent cycling, including:

   * Lower extremity fractures,
   * Severe joint contractures,
   * History of lower limb joint replacement,
   * Structural deformities of the lower extremities.
3. Severe communication, psychological, or psychiatric disorders (e.g., global aphasia) that impair the ability to follow instructions or complete assessments.
4. Participation in robot-assisted gait training or similar mechanically assisted rehabilitation interventions within the past 6 months prior to enrollment.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Quality | Baseline and 4 weeks
  Muscle quality will be assessed using the FITTO MQ device (Olive Healthcare, Seoul, Republic of Korea), which is based on discrete multi-wavelength near-infrared spectroscopy (DMW-NIRS). The device emits near-infrared light (650-1,100 nm) and analyzes reflected signals to estimate intramuscular composition, generating a muscle quality index (MQI).
  Measurements will be performed bilaterally at five muscle sites according to the standardized scan guide: erector spinae, rectus femoris, vastus lateralis, semitendinosus, and gastrocnemius. Each site will be measured twice on both the paretic and non-paretic sides, and the mean MQI value will be used for analysis. Higher MQI values indicate better muscle quality. Assessments will be conducted at baseline and after the 4-week intervention period.
Change in Fall Efficacy (K-FES-I) | Baseline and 4 weeks
  Falls efficacy will be evaluated using the Korean version of the Falls Efficacy Scale-International (K-FES-I). The K-FES-I is a validated self-reported questionnaire consisting of 16 items rated on a 4-point Likert scale, assessing concern about falling during daily activities.
  Although higher scores on the original scale indicate greater concern about falling, total scores will be reverse-coded for analysis in this study so that higher scores represent greater falls efficacy (i.e., less concern about falling and greater confidence during daily activities). The total score ranges from 16 to 64.
  Assessments will be conducted at baseline (Week 0) and after completion of the 4-week intervention (Week 4).
Change in Skeletal Muscle Mass Index (SMI) | Baseline and 4 weeks
  Skeletal muscle mass index (SMI) will be assessed using multi-frequency bioelectrical impedance analysis (BIA) with the ACCUNIQ BC720 system (T-SCAN PLUS III; SELVAS Healthcare, Seoul, Republic of Korea). This device applies electrical currents across a frequency range of 1-1,000 kHz to estimate whole-body and appendicular body composition, including skeletal muscle mass.
  Appendicular skeletal muscle mass (ASM) will be calculated as the sum of lean mass from both upper and lower extremities. SMI will be derived using the following formula:
  SMI (kg/m²) = ASM (kg) / height² (m²).
  Measurements will be conducted under standardized conditions with participants standing independently. Each participant will be measured twice, and the mean value will be used for analysis. Assessments will be performed at baseline and after the 4-week intervention period. Higher SMI values indicate greater skeletal muscle mass.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Score | Baseline and 4 weeks
  Physical function will be assessed using the electronic Short Physical Performance Battery (eSPPB; SPPB-100, Cybermedic Co., Seoul, Republic of Korea). The SPPB consists of three components: balance test (side-by-side, semi-tandem, and tandem stance), 4-meter gait speed test, and 5-times chair stand test. Each component is scored from 0 to 4 based on performance, yielding a total score ranging from 0 to 12, with higher scores indicating better physical performance.
  All assessments will be conducted by trained physical therapists with at least 3 years of clinical experience, who are blinded to group allocation. The eSPPB system incorporates infrared distance sensors, pressure sensors, and a balance platform to automatically detect task initiation and completion, thereby minimizing examiner-related timing errors and improving measurement reliability. Assessments will be performed at baseline and after the 4-week intervention period.
Change in Timed Up and Go Test (TUG) | Baseline and 4 weeks
  Functional mobility and dynamic balance will be assessed using the Timed Up and Go test (TUG). Participants will be instructed to rise from a chair with armrests, walk 3 meters at a comfortable pace, turn around, return to the chair, and sit down. The time required to complete the task will be recorded in seconds (to the nearest 0.1 s).
  Each participant will perform two trials using standardized verbal instructions, and the mean value will be used for analysis. Assessments will be conducted by trained physical therapists with at least 3 years of clinical experience. Testing will be discontinued if adverse events such as dizziness, pain, or unstable gait are observed. Lower TUG times indicate better functional mobility. Assessments will be performed at baseline and after the 4-week intervention period.
Change in Fugl-Meyer Assessment (FMA) Lower Extremity Score | Baseline and 4 weeks
  Lower extremity motor function will be assessed using the Fugl-Meyer Assessment for the Lower Extremity (FMA-LE), a standardized and widely used measure based on the neurological recovery framework for post-stroke motor impairment. The FMA-LE consists of 17 items scored on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully), yielding a total score ranging from 0 to 34, with higher scores indicating better voluntary motor control and coordination of the lower extremity.
  The assessment includes three subdomains: reflex activity, voluntary movement, and coordination/speed, covering selective movements of the hip, knee, and ankle. All assessments will be conducted by trained physical therapists with at least 3 years of clinical experience using standardized procedures. Assessments will be performed at baseline and after the 4-week intervention period.
Change in 6-Minute Walk Test (6MWT) | Baseline and 4 weeks
  Functional ambulation capacity and exercise tolerance will be assessed using the 6-Minute Walk Test (6MWT), conducted in accordance with the American Thoracic Society (ATS) guidelines. Participants will be instructed to walk as far as possible for 6 minutes at a self-selected pace, with the option to slow down or rest if needed. The total distance walked will be recorded in meters, with greater distances indicating better walking endurance and functional mobility.
  The test will be performed in a controlled indoor environment using a 40-meter rectangular loop track with a flat, non-elastic surface. Standardized verbal instructions and encouragement will be provided at 1-minute intervals. Participants may use their usual walking aids if required. The test will be discontinued immediately if adverse symptoms such as dizziness, chest pain, or severe fatigue occur. Assessments will be conducted at baseline and after the 4-week intervention period.
Change in Handgrip Strength | Baseline and 4 weeks
  Upper extremity muscle strength will be assessed using a digital handgrip dynamometer (TAKEI T.K.K.5401; Takei Scientific Instruments Co., Niigata, Japan). Measurements will be performed with participants seated, feet flat on the floor, shoulder in a neutral position, elbow flexed at 90°, and wrist in a neutral position. Handle span will be adjusted to fit each participant's hand size.
  Participants will be instructed to perform a maximal isometric contraction for 3-5 seconds. Two trials will be conducted for each hand, with a rest period of 30-60 seconds between trials to minimize fatigue. The maximum and mean values (kg) will be recorded for analysis. Lower grip strength values indicate reduced upper extremity muscle strength. Assessments will be conducted at baseline and after the 4-week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Seungwon Lee, PhD, Principal Investigator — Sahmyook University
Locations (1):
- Sahmyook University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the research team due to institutional policies and privacy regulations. Data will be securely stored and used solely for the purpose of this study and related publications.

REFERENCES:
- [Background] Gault ML, Willems ME. Aging, functional capacity and eccentric exercise training. Aging Dis. 2013 Sep 25;4(6):351-63. doi: 10.14336/AD.2013.0400351. PMID 24307968
- [Background] Iyanaga T, Abe H, Oka T, Miura T, Iwasaki R, Takase M, Isatake M, Doi A. Recumbent cycling with integrated volitional control electrical stimulation improves gait speed during the recovery stage in stroke patients. J Exerc Rehabil. 2019 Feb 25;15(1):95-102. doi: 10.12965/jer.1836500.250. eCollection 2019 Feb. PMID 30899743
- [Background] da Rosa Pinheiro DR, Cabeleira MEP, da Campo LA, Correa PS, Blauth AHEG, Cechetti F. Effects of aerobic cycling training on mobility and functionality of acute stroke subjects: A randomized clinical trial. NeuroRehabilitation. 2021;48(1):39-47. doi: 10.3233/NRE-201585. PMID 33386826
- [Background] Gonzalez-Rocha A, Mendez-Sanchez L, Ortiz-Rodriguez MA, Denova-Gutierrez E. Effect Of Exercise on Muscle Mass, Fat Mass, Bone Mass, Muscular Strength and Physical Performance in Community Dwelling Older Adults: Systematic Review and Meta-Analysis. Aging Dis. 2022 Oct 1;13(5):1421-1435. doi: 10.14336/AD.2022.0215. eCollection 2022 Oct 1. PMID 36186132
- [Background] Shin J, Park E. Comparison between Discrete Multi-Wavelength Near-Infrared Spectroscopy and Bioelectrical Impedance Analysis in the Assessment of Muscle Mass for Community-Dwelling Older People. J Clin Med. 2024 Apr 18;13(8):2350. doi: 10.3390/jcm13082350. PMID 38673621
- [Background] Menon RG, Raghavan P, Regatte RR. Quantifying muscle glycosaminoglycan levels in patients with post-stroke muscle stiffness using T1rho MRI. Sci Rep. 2019 Oct 10;9(1):14513. doi: 10.1038/s41598-019-50715-x. PMID 31601831
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Choi AY, Lim JH, Kim BG. Effects of muscle strength exercise on muscle mass and muscle strength in patients with stroke: a systematic review and meta-analysis. J Exerc Rehabil. 2024 Oct 25;20(5):146-157. doi: 10.12965/jer.2448428.214. eCollection 2024 Oct. PMID 39502116
- [Background] Hu MM, Wang S, Wu CQ, Li KP, Geng ZH, Xu GH, Dong L. Efficacy of robot-assisted gait training on lower extremity function in subacute stroke patients: a systematic review and meta-analysis. J Neuroeng Rehabil. 2024 Sep 19;21(1):165. doi: 10.1186/s12984-024-01463-1. PMID 39300491
- [Background] Calafiore D, Negrini F, Tottoli N, Ferraro F, Ozyemisci-Taskiran O, de Sire A. Efficacy of robotic exoskeleton for gait rehabilitation in patients with subacute stroke : a systematic review. Eur J Phys Rehabil Med. 2022 Feb;58(1):1-8. doi: 10.23736/S1973-9087.21.06846-5. Epub 2021 Jul 12. PMID 34247470
- [Background] Lorusso M, Tramontano M, Casciello M, Pece A, Smania N, Morone G, Tamburella F. Efficacy of Overground Robotic Gait Training on Balance in Stroke Survivors: A Systematic Review and Meta-Analysis. Brain Sci. 2022 May 31;12(6):713. doi: 10.3390/brainsci12060713. PMID 35741599
- [Background] Su Y, Yuki M, Otsuki M. Prevalence of stroke-related sarcopenia: A systematic review and meta-analysis. J Stroke Cerebrovasc Dis. 2020 Sep;29(9):105092. doi: 10.1016/j.jstrokecerebrovasdis.2020.105092. Epub 2020 Jul 3. PMID 32807486
- [Background] Louie DR, Mortenson WB, Durocher M, Teasell R, Yao J, Eng JJ. Exoskeleton for post-stroke recovery of ambulation (ExStRA): study protocol for a mixed-methods study investigating the efficacy and acceptance of an exoskeleton-based physical therapy program during stroke inpatient rehabilitation. BMC Neurol. 2020 Jan 28;20(1):35. doi: 10.1186/s12883-020-1617-7. PMID 31992219
- [Result] Scherbakov N, Doehner W. Sarcopenia in stroke-facts and numbers on muscle loss accounting for disability after stroke. J Cachexia Sarcopenia Muscle. 2011 Mar;2(1):5-8. doi: 10.1007/s13539-011-0024-8. Epub 2011 Mar 25. PMID 21475676